CLINICAL TRIAL: NCT04228796
Title: Analysis of Biomarkers in Lymph Node Tissue
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Other Study IDs: 19-011883
Record Dates: First submitted 2020-01-11; First posted 2020-01-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Analysis of Biomarkers in Lymph Node Tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are doing an exploratory analysis of biomarkers to correlate with treatment outcome of transplant surgery.

DETAILED DESCRIPTION:
Researchers will study previously collected tissue, which was sent for pathological examination, of 200 patients who underwent transplant surgery. Concentration of biomarkers in lymph node tissue will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+years of age)
* Undergo any organ transplant

Exclusion Criteria:

* Under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Analysis will be done on previously collected tissue of 200 adult subjects who underwent transplant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
List of biomarkers | Baseline
  Immunohistochemistry (IHC) for the LYVE1, VEGFR3 expression, VEGF-A/C/D, Ki-67, MMP-9 and TIMP-1

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials